CLINICAL TRIAL: NCT05929742
Title: The Efficacy of Early Rehabilitation Combined With Virtual Reality Training in Patients With First-time Acute Stroke
Brief Title: Early Rehab With VR for First-time Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Ta-Chung Chao, Doctor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001-VR
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute; Acute Ischemic Stroke
Keywords: Early rehabilitation; Virtual reality
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups: the experimental group, which received early rehabilitation combined with VR training, and the comparison group, which received only early rehabilitation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): received early rehabilitation combined with VR training
  Interventions: Behavioral: virtual reality training; Behavioral: early rehabilitation
- comparison group (Active Comparator): received only early rehabilitation
  Interventions: Behavioral: early rehabilitation

INTERVENTIONS:
Behavioral: virtual reality training — The experimental group received five additional days of supervised VR training using a wireless sensor in a private room in the neurological care ward.
  Arms: experimental group
Behavioral: early rehabilitation — Five 60-minute sessions per week, was prescribed by a rehabilitation physician and performed by physical, occupational, and speech therapists from 3 to 6 days after admission.

SUMMARY:
The goal of this clinical trial is to confirm the efficacy and feasibility of early rehabilitation combined with virtual reality training in patients following first-time acute stroke. The main questions it aims to answer are:

* The impact of virtual reality training on muscle strength;
* The impact of virtual reality training on functional recovery;
* The impact of virtual reality training on mood state.

Researchers will compare the experimental group, which received early rehabilitation combined with VR training, and the comparison group, which received only early rehabilitation, to see if VR training has clinical benefits when provided alongside early rehabilitation during hospitalization.

DETAILED DESCRIPTION:
Early rehabilitation has been shown to enhance outcomes for patients with first-time acute stroke. However, whether the addition of virtual reality (VR) training could further improve muscle strength, functional recovery, and mood state for these patients is unknown. Therefore, this study aimed to investigate the effectiveness of early rehabilitation combined with VR training in patients following first-time acute stroke. Patients with acute ischemic stroke will be selected and randomly assigned with a 1:1 randomization ratio to either the experimental group or the comparison group. Both groups received early rehabilitation, and the experimental group received extra VR training starting 24 hours to 3 days poststroke during the stay in the hospital. Muscle strength, functional status, and mood state will be collected before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* first-time acute infarction (ischemic stroke);
* admission to the hospital within three days of stroke onset;
* able to communicate with verbal or nonverbal methods and understand Mandarin;
* had a disability that ranged from minimal to moderately severe disability and evaluated as 1-4 scores by the modified Rankin Scale (mRS);
* agree to be randomized.

Exclusion Criteria:

* diagnosis of global aphasia, transient ischemic attack, visual or auditory impairment;
* mRS over 5 (severe disability: requires constant nursing care and attention, bedridden, incontinent);
* a history of cancer, end-stage renal disease with dialysis, dementia, mental health disorders (particularly major depression), based on both of medical records and assessments from the neurologist;
* being unable to participate due to other comorbid neurological and musculoskeletal conditions that produce moderate-to-severe physical disability;
* prolonged stay in hospital for over three weeks due to other medical diseases (e.g., myocardial infarction, septic shock, cancer) after admission or length of stay in hospital less than one week due to a decline to treatment and transferred to another hospital for further confirmation of diagnosis and other complementary or alternative therapies.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-08-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
muscle strength | through the admission period, an average of 1 month
  The testing involved assessing the patient's upper and lower limb/extremities muscles against the examiner's resistance and grading the patient's strength on a 0-5 scale, higher scores mean a better outcome.
postural control | through the admission period, an average of 1 month
  The Postural Assessment Scale for Stroke (PASS), consisting of two sections with a 4-point scale, with 0 being the lowest level of functionality and 3 the highest, and a total score ranging from 0-36, is a well-validated clinical assessment tool for postural control in patients with stroke during the first three months after stroke.
activities of daily living | through the admission period, an average of 1 month
  The Barthel scale used to assess individuals' performance in activities of daily living has high inter-rater reliability and test-retest reliability as well as high correlations with other measures of physical disability. The scores of the 10-item Barthel scale range from 0-100 with 5-point increments. Patients with higher scores are more independent than those with lower scores in their daily activities.
mood state | through the admission period, an average of 1 month
  Mood state was assessed by the Hospital Anxiety and Depression Scale (HADS). This well-validated tool has 14 items (7 items related to anxiety [HADS-A] and 7 related to depression [HADS-D]). Each item of the HADS is scored from 0-3, and the range is 0-21 for depression and anxiety. Participants with higher scores represent a higher level of depression or anxiety. A cut-off point of 8 has been identified for anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Lin Chiang, MD, PHD, Study Director — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no intention to share the individual participant data (IPD) collected in this study with other researchers. This decision was influenced by factors such as privacy concerns, confidentiality agreements, legal restrictions, institutional policies that restrict the sharing of sensitive or proprietary data, and ethical considerations to protect the privacy and confidentiality of the participants involved in the study. Therefore, the data will be kept from other researchers.

REFERENCES:
- [Background] Khan A, Podlasek A, Somaa F. Virtual reality in post-stroke neurorehabilitation - a systematic review and meta-analysis. Top Stroke Rehabil. 2023 Jan;30(1):53-72. doi: 10.1080/10749357.2021.1990468. Epub 2021 Nov 7. PMID 34747351
- [Background] Hao J, Yao Z, Harp K, Gwon DY, Chen Z, Siu KC. Effects of virtual reality in the early-stage stroke rehabilitation: A systematic review and meta-analysis of randomized controlled trials. Physiother Theory Pract. 2023 Dec 2;39(12):2569-2588. doi: 10.1080/09593985.2022.2094302. Epub 2022 Jul 7. PMID 35801290
- [Background] da Silva Cameirao M, Bermudez I Badia S, Duarte E, Verschure PF. Virtual reality based rehabilitation speeds up functional recovery of the upper extremities after stroke: a randomized controlled pilot study in the acute phase of stroke using the rehabilitation gaming system. Restor Neurol Neurosci. 2011;29(5):287-98. doi: 10.3233/RNN-2011-0599. PMID 21697589
- [Background] Lee SJ, Chun MH. Combination transcranial direct current stimulation and virtual reality therapy for upper extremity training in patients with subacute stroke. Arch Phys Med Rehabil. 2014 Mar;95(3):431-8. doi: 10.1016/j.apmr.2013.10.027. Epub 2013 Nov 14. PMID 24239790
- [Background] Chen L, Lo WL, Mao YR, Ding MH, Lin Q, Li H, Zhao JL, Xu ZQ, Bian RH, Huang DF. Effect of Virtual Reality on Postural and Balance Control in Patients with Stroke: A Systematic Literature Review. Biomed Res Int. 2016;2016:7309272. doi: 10.1155/2016/7309272. Epub 2016 Dec 7. PMID 28053988
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493